CLINICAL TRIAL: NCT04863183
Title: Cell Therapy for Patients With Symptomatic Knee Osteoarthritis: Phase I / II, Controlled, Randomized and Double-blind Clinical Trial
Brief Title: Cell Therapy With Cellistem-OA for Symptomatic Knee Osteoarthritis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundación Oftalmológica de Santander Clínica Carlos Ardila Lulle (Other)
Collaborators: Cells for Cells (Industry)
Responsible Party: Principal Investigator, Martha Ligia Arango Rodríguez, Director Technical and Scientific Centro de Terapias Avanzadas Fundación Ofalmológica de Santander, Fundación Oftalmológica de Santander Clínica Carlos Ardila Lulle
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OA-01
Record Dates: First submitted 2021-04-20; First posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Mesenchymal Stem Cells; Knee Osteoarthritis; Cell Therapy
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Triamcinolone Acetonide; Triamcinolone

STUDY DESIGN:
Intervention Model Description: Controlled, randomized, double-blind clinical trial comparing CELLISTEM-OA and active comparator (triamcinolone acetonide).
Who Masked: Participant, Care Provider, Investigator
Masking Description: The Center for Advanced Therapies will send a pre-filled syringe with the 5 cc of solution without any difference in its external appearance, regardless of the content, according to the previously randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (control-Triamcinolone acetonide) (Active Comparator): Triamcinolone acetonide (10mg / mL) via intra-articular, 5 cc, one dose (zero time).
  Interventions: Drug: Triamcinolone acetonide
- Group 2 (experimental- CELLISTEM-OA) (Experimental): CELLISTEM-OA via intra-articular, doses of 2 x 106 mesenchymal stem cells in 5cc of saline solution, one dose (zero time).
  Interventions: Biological: CELLISTEM-OA

INTERVENTIONS:
Biological: CELLISTEM-OA — The intra-articular puncture will be performed by an orthopedic doctor specializing in knee and hip treatments. The procedure will be carried out using sterile technique, after cooling the skin with local ice.
  Other Names: Mesenchymal stem cells
  Arms: Group 2 (experimental- CELLISTEM-OA)
Drug: Triamcinolone acetonide — The intra-articular puncture will be performed by an orthopedic doctor specializing in knee and hip treatments. The procedure will be carried out using sterile technique, after cooling the skin with local ice.
  Other Names: Kenacort-A
  Arms: Group 1 (control-Triamcinolone acetonide)

SUMMARY:
Symptomatic knee osteoarthritis is a serious public health problem in the world, it carries a high personal, social and economic impact. Currently, there are no drugs that modify the natural course of the disease. As analgesic therapy becomes insufficient, more invasive measures are applied, ultimately leading to arthroplasty.

The scientific community has joined efforts to develop new therapeutic approaches that allow the delay and regeneration of injured tissue in these patients. These include cell therapy with mesenchymal stem cells derived from different sources. Although most of the clinical studies carried out in different parts of the world with this therapy in patients with knee osteoarthritis have shown therapeutic benefit, it is necessary to develop clinical trials with high quality in our population.

The aim of this project is to evaluate the safety, tolerance and efficacy of Cellistem-OA (biological therapy based on mesenchymal stem cells derived from Wharton's jelly of umbilical cord) in patients with knee osteoarthritis in the Colombian population.

Investigators proposed to carry out an experimental (clinical trial), randomized, controlled and parallel with 30 participants with knee knee osteoarthritis of the medical complex Fundación Oftalmológica de Santander Clínica Carlos Ardila Lulle. The participants will be randomized into two groups: i) 15 patients who will receive a dose of 2 x 106 Cellistem-OA and ii) 15 patients who will receive an active comparator (acetonide of triamcinolone 10mg / mL), which will be administered by intra-articular injection in the superolateral aspect of the knee. The outcomes to be evaluated will be: (i) decrease in joint pain, (ii) increase in joint functionality, (iii) improvement in quality of life and (iv) improvement of articular cartilage. These parameters will be evaluated at weeks 1, 4, 8, 12, 24, 25, 28, 32, 36 and 52 post-treatments. Additionally, local and systemic adverse events will be recorded to establish whether or not there is an association between them and the intervention.

DETAILED DESCRIPTION:
Type of study Controlled, randomized, double-blind clinical trial comparing CELLISTEM-OA and active comparator (triamcinolone acetonide).

Study population Patients from the Fundación Oftalmológica de Santander Clínica Carlos Ardila Lulle who consult the trauma and rheumatology service by knee osteoarthritis. Patients who show interest in participating will be cited to an interview with the researchers where both the objectives and the research procedures will be explained.

Sample size The sample size considered are 30 participants distributed in two groups.

Group 1 (control) active comparator: triamcinolone acetonide (10mg / mL) via intra-articular, 5 cc.

Group 2 (experimental): CELLISTEM-OA via intra-articular, doses of 2 x 106 cells in 5cc of saline solution.

The intra-articular puncture will be performed by an orthopedic doctor specializing in knee and hip treatments using sterile technique, after cooling the skin with local ice.

ELIGIBILITY:
Inclusion Criteria:

Patients who / with:

* Osteoarthritis of the knee.
* Kellgren II or III to knee radiography.
* 30 to 75 years inclusive.
* Pain scale greater than 40 over 100 mm.
* MRI with G I, II or III chondral knee injury with or without stable degenerative meniscal injury.
* Stable knee.
* Examination of the rest of the normal limb.
* Willingness to participate in the study for 1 year.
* Ability to understand and willingness to sign the informed consent.

Exclusion Criteria:

Patients who / with:

* Symptomatic contralateral knee osteoarthritis.
* Significant knee trauma in the preceding 3 months.
* Wound or skin lesion in the knee studied.
* Anatomical valgus greater than 10º.
* Anatomical varus greater than 5º.
* Clinically significant joint effusion.
* Edema greater than 20% of the surface of the plateau or condyle in NMR.
* Previously known alterations in the hip and / or spine.
* Predominant patellofemoral pathology (radiographs with IWANO II osteoarthritis or more).
* Any type of inflammatory arthritis.
* History of active infections including HIV, HBV and HCV.
* Results of laboratory tests (hemogram and CRP) outside the normal ranges.
* Presence of fever on day -1 or day 0.
* Use of oral corticosteroids.
* Use of anticoagulants.
* Immunosuppression, uncontrolled diabetes mellitus, hyperthyroidism, psychiatric illnesses
* Active neoplasia or during the preceding 5 years.
* Pregnancy or breastfeeding (b-Hcg positive).
* Use of drugs or alcoholism.
* IA injections or knee surgeries in the last 180 days.
* BMI> 35.
* Any type of metallic implant susceptible to displacement with MRI.
* Use of pacemakers.
* History of severe allergy or anaphylactic shock.
* Significant alterations in the evaluation of the initial laboratory tests.
* Any factor that, in the opinion of the investigator, may affect the adequate follow-up of the patient during the study

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Decrease in joint pain | 12 months
  Pain will be measured through visual analog scale (VAS).
Increased joint functionality | 12 months
  Joint functionality will be measured through the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC).
Improvement in the quality of life | 12 months
  Quality of life will be measured through the Short Form 36 Health Survey Questionnaire (SF-36).
Imaging improvement of articular cartilage | 12 months
  The improvement of articular cartilage will be evaluated by nuclear magnetic resonance (NMR).

CONTACTS AND LOCATIONS:
Overall Officials: Martha L Arango, PhD, Principal Investigator — Fundación Oftalmológica de Santander Clínica Carlos Ardila Lulle

IPD SHARING:
Plan to Share IPD: No